CLINICAL TRIAL: NCT03261011
Title: A Phase 1A/1B Multicenter, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK104 in Subjects With Advanced Solid Tumors
Brief Title: Study of the Safety, Pharmacokinetics, and Antitumor Activity of AK104 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-101
Record Dates: First submitted 2017-08-20; First posted 2017-08-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cancer
Keywords: immunotherapy; immuno-oncology; advanced solid tumors

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK-104 (Experimental): Single-arm
  Interventions: Biological: AK-104

INTERVENTIONS:
Biological: AK-104 — Subjects will receive AK104 by intravenous administration.

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of AK104 as a single agent in adult subjects with advanced solid tumor malignancies. The study consists of a dose escalation phase (Phase 1a) to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for AK104 as a single agent, and a dose expansion phase (Phase 1b) which will characterize treatment of AK104 as a single agent at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent and any locally required authorization obtained from the subject/legal representative.
* In dose-escalation cohorts (Phase 1a), histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
* In the dose-expansion cohorts (Phase 1b), histologically or cytologically confirmed selected advanced solid tumors (to be determined). Subjects must have received no more than three prior lines of systemic therapy for advanced or metastatic disease.
* Subject must have at least one measurable lesion according to RECIST Version1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
* Available archived tumor tissue sample to allow for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use, the subject must consent and undergo fresh tumor biopsy.
* Adequate organ function.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTL4 antibody or any other antibody or drug targeting T-cell costimulation or checkpoint pathways such as ICOS, or agonists such as CD40, CD137, GITR, OX40 etc.
* Receipt of any immunotherapy, any conventional or investigational systemic anticancer therapy within 4 weeks prior to the first dose of AK104; in the case of mAbs, 6 weeks prior to the first dose of AK104.
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions is acceptable.
* Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
* Active or prior documented autoimmune disease within the past 2 years.
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplant or hematopoietic stem cell that requires use of immunosuppressives.
* Known allergy or reaction to any component of the AK104 formulation.
* History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
* Known history of tuberculosis.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection except for subjects with HCC.
* An active infection requiring systemic therapy with the exception of anti-viral therapy for hepatitis as specified by the protocol.
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of AK104.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of AK104, up to 2 years and 3 months
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 4 weeks
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 3 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | Up to 3 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 3 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 3 years
  Overall survival is defined as the time from the start of treatment with AK104 until death due to any cause.
Area under the curve (AUC) of AK104 | From first dose of AK104 through 90 days after last dose of AK104; Up to 2 years and 3 months.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Maximum observed concentration (Cmax) of AK104 | From first dose of AK104 through to 90 days after last dose of AK104; Up to 2 years and 3 months.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of AK104 through to 90 days after last dose of AK104; Up to 2 years and 3 months.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through to 90 days after last dose of AK104; Up to 2 years and 3 months.
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Integrated Clinical Oncology Network (ICON), South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research/Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Li X, Xiao G, Desai J, Frentzas S, Wang ZM, Xia Y, Li B. CD74 is associated with inflamed tumor immune microenvironment and predicts responsiveness to PD-1/CTLA-4 bispecific antibody in patients with solid tumors. Cancer Immunol Immunother. 2024 Jan 27;73(2):36. doi: 10.1007/s00262-023-03604-2. PMID 38280003
- [Derived] Frentzas S, Gan HK, Cosman R, Coward J, Tran B, Millward M, Zhou Y, Wang W, Xia D, Wang ZM, Li B, Xia M, Desai J. A phase 1a/1b first-in-human study (COMPASSION-01) evaluating cadonilimab in patients with advanced solid tumors. Cell Rep Med. 2023 Nov 21;4(11):101242. doi: 10.1016/j.xcrm.2023.101242. Epub 2023 Oct 17. PMID 37852261
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37852261/